CLINICAL TRIAL: NCT03127956
Title: An Open-Label Study Assessing Long-Term Safety of Olumacostat Glasaretil Gel in Subjects With Acne Vulgaris
Brief Title: A Long-term Safety Study of Olumacostat Glasaretil Gel in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRM01B-ACN05
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Results first posted 2019-02-05 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olumacostat Glasaretil Gel, 5.0% (Experimental): Olumacostat Glasaretil Gel, 5.0%, applied twice daily to the face
  Interventions: Drug: Olumacostat Glasaretil Gel, 5.0%

INTERVENTIONS:
Drug: Olumacostat Glasaretil Gel, 5.0% — Gel containing Olumacostat Glasaretil
  Other Names: DRM01B

SUMMARY:
The objective of this study is to assess the long-term safety of Olumacostat Glasaretil gel, 5.0% in patients with acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent or assent (for subjects under legal adult age)
* Completed Week 12 visit of either DRM01B-ACN03 or DRM01B-ACN04 studies.
* Willing to comply with the protocol. Subjects under legal adult age will be assessed by the investigator as to their ability to comply with the protocol
* Willing to refrain from using any treatments on the face for acne vulgaris, other than the investigational product, including topical or systemic antibiotics.

Exclusion Criteria:

* Abnormal clinically significant findings on physical exam, vital signs or ECG at Week 12 visit of either the DRM01-ACN03 or DMR01-ACN04 studies that would make further treatment with Olumacostat Glasaretil Gel contraindicated, as determined by the Investigator
* Any other condition which, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 748 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Zib, Study Director — Dermira, Inc.
Locations (94):
- United States (73):
  - Avant Research Associates, LLC, Guntersville, Alabama
  - Advanced Research Associates, Glendale, Arizona
  - Alliance Dermatology & MOHS Center, Phoenix, Arizona
  - Dermatology Trial Associates, Bryant, Arkansas
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Anaheim Clinical Trials, Anaheim, California
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Advanced Skincare Surgery & MedCenter, Fullerton, California
  - Dermatology Research Associates, Los Angeles, California
  - Northern California Research, Sacramento, California
  - Rady Children's Hospital UCSD Pediatric and Adolescent Derm, San Diego, California
  - TCR Medical Corporation, San Diego, California
  - University Clinical Trials Inc., San Diego, California
  - Radiant Research, Inc., Santa Rosa, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Horizons Clinical Research Center, LLC, Denver, Colorado
  - Dermatology Physicians of CT, Shelton, Connecticut
  - Center for Clincial and Cosmetic Research, Aventura, Florida
  - Florida Academic Centers Research & Education, Coral Gables, Florida
  - Aby's New Generation Research Inc., Hialeah, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Finlay Medical Research, Miami, Florida
  - Floridian Research Institute, Miami, Florida
  - Pioneer Clinical Research, Pembroke Pines, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Health Awareness, Inc, Port Saint Lucie, Florida
  - International Clinical Research-US, LLC, Sanford, Florida
  - Lenus Research & Medical Group, Sweetwater, Florida
  - MOORE Clinical Research, Inc, Tampa, Florida
  - Visions Clinical Research, Wellington, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Marietta Dermatology Clinical Research, Inc., Marietta, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Forefront Dermatology, Carmel, Indiana
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Skin Sciences, PLLC, Louisville, Kentucky
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Lawrence Jeffrey Green MD, LLC, Rockville, Maryland
  - Great Lakes Research Group, Inc, Bay City, Michigan
  - Henry Ford Medical Center, New Center One, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Mercy Research, Washington, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Quality Clinical Research Inc., Omaha, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - JDR Dermatology Research, LLC, Las Vegas, Nevada
  - Acne Treatment & Research Center, Morristown, New Jersey
  - Schweiger Dermatology, PLLC, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - DermResearchCenter of New York, Inc., Stony Brook, New York
  - Sterling Research Group, Cincinnati, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Meridian Clincial Research, Dakota Dunes, South Dakota
  - The Skin Wellness Center, Knoxville, Tennessee
  - International Clinical Research - Tennessee LLC, Murfreesboro, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch, Inc, Austin, Texas
  - Avant Research Associates, Beaumont, Texas
  - J&S Studies, Inc., College Station, Texas
  - Synexus US, LP, dba, Research Across America, Dallas, Texas
  - Suzanne Bruce and Associates, P.A. The Center for Skin Research, Houston, Texas
  - Austin Institute for Clinical Research, Inc, Pflugerville, Texas
  - Synexus US, LP, dba, Research Across America, Plano, Texas
  - Progressive Clinical Research, PA, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Dermatology Clinical Research Center of San Antonio, San Antonio, Texas
  - Houston Center for Clinical Research, Sugar Land, Texas
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Premier Clinical Research, Spokane, Washington
- Australia (10):
  - Woden Dermatology, Phillip, Australian Capital Territory
  - Premier Specialists, Kogarah, New South Wales
  - St George Dermatology and Skin Cancer Centre, Kogarah, New South Wales
  - The Skin Centre, Benowa, Queensland
  - Veracity Clinical Research, Woolloongabba, Queensland
  - North Eastern Health Specialists, Hectorville, South Australia
  - Skin & Cancer Foundation Inc., Carlton, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Fremantle Dermatology, Fremantle, Western Australia
  - Burswood Dermatology, Victoria Park, Western Australia
- Canada (11):
  - Institute for Skin Advancement, Calgary, Alberta
  - Enverus Medical Research, Surrey, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology Center, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - XLR8 Medical Research, Windsor, Ontario
  - Windsor Research Inc., Windsor, Ontario

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Olumacostat Glasaretil Gel, 5.0%
Started | 748
Completed | 431
Not Completed | 317

BASELINE CHARACTERISTICS:
Population: The Total Participants at risk are based on the Safety population, defined as, Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Olumacostat Glasaretil Gel, 5.0%
Number analyzed (Participants) | 741
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 446
  Between 18 and 65 years | 295
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 19.3 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 423
  Male | 318
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 211
  Not Hispanic or Latino | 522
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 26
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 133
  White | 546
  More than one race | 29
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 30
  United States | 625
  Australia | 86

OUTCOME MEASURES:

1. Primary Outcome: Long-Term Safety Assessed Through Adverse Events and Local Skin Reactions
Description: Long-Term Safety Assessed Through Adverse Events and Local Skin Reactions
Time Frame: Day 1 - Week 36
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Olumacostat Glasaretil Gel, 5.0%
Number analyzed (Participants) | 741
Participants
  Adverse Events (Mild) | 197
  Adverse Events (Moderate) | 124
  Adverse Events (Severe) | 18
  Adverse Events (Not Reported) | 402
  Burning/Stinging (None) | 518
  Burning/Stinging (Mild) | 11
  Burning/Stinging (Moderate) | 2
  Burning/Stinging (Severe) | 0
  Burning/Stinging (Not Reported) | 210
  Pruritus (None) | 500
  Pruritus (Mild) | 29
  Pruritus (Moderate) | 2
  Pruritus (Severe) | 0
  Pruritus (Not Reported) | 210
  Erythema (None) | 469
  Erythema (Mild) | 55
  Erythema (Moderate) | 7
  Erythema (Severe) | 0
  Erythema (Not Reported) | 210
  Dryness (None) | 485
  Dryness (Mild) | 43
  Dryness (Moderate) | 3
  Dryness (Severe) | 0
  Dryness (Not Reported) | 210
  Peeling (None) | 507
  Peeling (Mild) | 22
  Peeling (Moderate) | 1
  Peeling (Severe) | 0
  Peeling (Not Reported) | 211

ADVERSE EVENTS:
Time Frame: Baseline to Week 36
Description: The Total Participants at risk are based on the Safety Population defined as Participants who were randomized and received at least one confirmed dose of study drug.
Arm/Group | Olumacostat Glasaretil Gel, 5.0%
All-Cause Mortality (participants affected / at risk) | 0/741
Serious Adverse Events (participants affected / at risk) | 8/741
Other Adverse Events (participants affected / at risk) | 281/741
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 5.0% (N=741)
Infectious mononucleosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Epilepsy (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olumacostat Glasaretil Gel, 5.0% (N=741)
Application site dryness (General disorders) | 28
Application site erythema (General disorders) | 25
Application site pain (General disorders) | 29
Application site pruritus (General disorders) | 39
Influenza (Infections and infestations) | 16
Nasopharyngitis (Infections and infestations) | 49
Upper respiratory tract infection (Infections and infestations) | 57
Sunburn (Injury, poisoning and procedural complications) | 19
Headache (Nervous system disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT03127956/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT03127956/SAP_001.pdf